CLINICAL TRIAL: NCT06450769
Title: Effect of Mediterranean Diet Supplemented With Aronia and Low-Fat Diet on Hepatic Steatosis, Inflammation, Oxidative Stress and Microbiota in Non-alcoholic Fatty Liver Disease
Brief Title: Aronia and Non-alcoholic Fatty Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Kent University (Other)
Responsible Party: Principal Investigator, Gamze Akbulut, Professor Doctor, Istanbul Kent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 222S452
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Aronia; NAFLD; Mediterranean diet; Oxidative stress; Inflammation; Microbiota
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Inflammation | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mediterranean diet group (Experimental): An individually planned nutrition program suitable for the energy-restricted Mediterranean diet will be created for individuals in this group.
  Interventions: Other: Mediterranean diet
- Mediterranean diet supplemented with aronia group (Experimental): An individually planned nutrition program suitable for the energy-restricted Mediterranean diet will be created for individuals in this group. Also 100 mL/day of 100% aronia juice will be given.
  Interventions: Other: Aronia juice; Other: Mediterranean diet
- Low-fat diet group (Experimental): An individually planned nutrition program suitable for the energy-restricted low-fat diet will be created for individuals in this group.
  Interventions: Other: Low-fat diet
- Low-fat diet supplemented with aronia group (Experimental): An individually planned nutrition program suitable for the energy-restricted low-fat diet will be created for individuals in this group. Also 100 mL/day of 100% aronia juice will be given.
  Interventions: Other: Aronia juice; Other: Low-fat diet

INTERVENTIONS:
Other: Aronia juice — 100% aronia juice, 100 mL/day, twelve-week follow-up
  Arms: Low-fat diet supplemented with aronia group; Mediterranean diet supplemented with aronia group
Other: Mediterranean diet — An individually planned nutrition program suitable for the energy-restricted Mediterranean diet
  Arms: Mediterranean diet group; Mediterranean diet supplemented with aronia group
Other: Low-fat diet — An individually planned nutrition program suitable for the energy-restricted low-fat diet
  Arms: Low-fat diet group; Low-fat diet supplemented with aronia group

SUMMARY:
Adults newly diagnosed with NAFLD will be included in the study. At the beginning of the research, the socio-demographic characteristics and nutritional habits of the individuals will be questioned with a face-to-face questionnaire. In addition, at the beginning of the study, blood samples, 3-day food consumption record, physical activity record, anthropometric measurements (height, body weight, waist, hip and neck circumference and body composition analysis) and stool samples will be taken from the patients. Oxidative stress (TAS, TOS, SOD, Malondialdehyde, Catalase, Glutathione peroxidase, Glutathione, AGE and DNA oxidative damage) and inflammation (CRP, TNF-alpha, IL-17, IL-23, IL-10, IL-13, TGF-beta) parameters in blood samples will be analyzed. Patients will then be randomized into four groups to follow a Mediterranean diet supplemented with aronia, a Mediterranean diet, a low-fat diet supplemented with aronia, or a low-fat diet. Necessary training will be given to the participants so that they can apply the individually planned diet. Dietary adherence and anthropometric measurements will be evaluated every 2 weeks. At the end of the twelve-week follow-up, all parameters evaluated at the beginning of the study will be repeated and compared with previous values.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a chronic liver disease in which more than 5% fat accumulation in the liver (steatosis). It has become the most common liver disease in adults with the effect of obesity. In fact, NAFLD is seen in approximately 25% of adults. If left untreated, it can progress to cirrhosis, hepatocellular carcinoma, and end-stage liver failure. It is obvious that it is necessary to identify preventive factors for NAFLD and to develop new approaches for its treatment. There is an increase in inflammation and oxidative stress levels in NAFLD, which is important for the development of possible treatment methods. In this study, the Mediterranean diet supplemented with aronia is expected to contribute positively to progression of the disease by improving inflammation and oxidative stress parameters. Adding aronia to the Mediterranean diet will increase the polyphenol content of this diet. This study was planned with the thought that a Mediterranean diet supplemented with aronia will have positive effects on hepatic steatosis, oxidative stress, inflammation, and microbiota in NAFLD, where lifestyle changes, including healthy nutrition, are included in the primary treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18- 64 years of age
* Body mass index (BMI) 25-40 kg/m2
* Newly diagnosed with NAFLD and has not been treated before
* Volunteering

Exclusion Criteria:

* Chronic disease other than NAFLD
* Pregnancy or breastfeeding
* Bleeding disorder
* Regular medication use
* Any food allergies or intolerances
* Being on a special diet treatment
* Smoking in the last year
* Alcohol use in the last year
* Having used antibiotics in the last 3 months
* Use of prebiotics or probiotics in the last 3 months
* Use of proton pump inhibitors in the last 3 months
* Use of vitamin-mineral supplementation in the last 3 months
* Use of nutritional supplements in the last 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress | Baseline and end of the 12th week
  TAS, TOS, SOD, Malondialdehyde (MDA), Catalase, Glutathione peroxidase, Glutathione, AGE and DNA oxidative damage will be evaluated.
Inflammation | Baseline and end of the 12th week
  CRP, TNF-alfa, IL-10, IL-13, IL-17, IL-23, TGF-β, LPS will be evaluated.
Degree of hepatic steatosis | Baseline and end of the 12th week
  Evaluation of hepatic steatosis by liver ultrasonography
Microbiota analysis | Baseline and end of the 12th week
  16s rRNA Gene Sequencing and Compositional Analyzes
Body composition analysis | Baseline, every 15 days and end of the 12th week
  Body weight, height and body composition, waist, hip and neck circumference measurements

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Akbulut, Study Director — Kent University; Tarkan Karakan, Principal Investigator — Gazi University; Ali Karataş, Principal Investigator — Gazi University; Emine Yassıbaş, Principal Investigator — Gazi University; Feride Ayyıldız, Principal Investigator — Gazi University; Büşra Atabilen, Principal Investigator — Karamanoğlu Mehmetbey University

IPD SHARING:
Plan to Share IPD: No